CLINICAL TRIAL: NCT05648461
Title: The Accelerate Trial: Phase II Study Exploring Five Fractions of Accelerated Hypofractionated Post-operative Radiation Therapy in Head and Neck Cancer
Brief Title: Phase II Study Exploring Five Fractions of Post-operative Radiation Therapy in Head and Neck Cancer
Acronym: Accelerate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aman Sharma, Aman Sharma, All India Institute of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: The Accelerate Trial
Record Dates: First submitted 2022-12-04; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Five fraction of post operative Radiotherapy (Experimental): The present study is a non -randomised phase II study that will enroll 50 patients and test feasibility of 30 Gy in 5 fractions of the primary disease and ipsilateral level I-III disease.
  Interventions: Radiation: Five fraction of post operative radiotherapy

INTERVENTIONS:
Radiation: Five fraction of post operative radiotherapy — Target volume will include tumor bed & ipsilateral level I-III levels.

SUMMARY:
The purpose of this research study is to investigate a shorter radiation treatment schedule for head and neck cancers. The present study is a non -randomized phase II study that will enroll 50 patients and test feasibility of 30 Gy in 5 fractions of the primary disease and ipsilateral level I-III disease.

DETAILED DESCRIPTION:
Radiotherapy (RT) is an integral cancer treatment and RT utilization rates for commonly occurring carcinoma include breast: 87%, cervical: 71%, head and neck: 84%, lung: 77%, and prostate: 58% [1]. Overall, 57.5% of global head and neck cancers occur in Asia especially in India [2]. Head and neck cancers in India accounted for 30% of all cancers. In India, 60 to 80% of patients present with advanced disease as compared to 40% in developed countries [3]. Inequitable radiotherapy availability in India leads to non-compliance in many cases, as patients need to travel long distances for treatment. The number of functional radiotherapy units in India is below the limit recommended by the World Health Organization [3]. This poses a serious barrier to radiotherapy access as well as timely delivery of multidisciplinary cancer care.

Post operative radiation treatment for head and neck patients requires 6 weeks of time and the patient has to travel to the radiotherapy department daily for 5 days a week. This long course of radiation can lead to significant side effects resulting in some people being unable to complete the course of treatment. The Accelerate trial has potential to provide a quick solution (by reducing 30 fractions of PORT to 5 fractions) and is particularly suitable for resource constraint and overburdened radiotherapy. Five fractions of radiotherapy has been proven to be equally efficacious to long courses at various cancer sites like rectal cancer, breast cancer [4,5]. With small volume disease and technological advances in delivery of radiotherapy it is possible to deliver 5 fractions of hypofractionated RT to prostate, lung and pancreatic cancer [6-8].

The present study is a non -randomised phase II study that will enroll 50 patients and test feasibility of 30 Gy in 5 fractions of the primary disease and ipsilateral level I-III disease.

References

1. Atun R, Jaffray DA, Barton MB, et al: Expanding global access to radiotherapy. Lancet Oncol 16:1153-1186, 2015.
2. Chaturvedi P. Head and neck surgery. J Can Res Ther 2009; 5:143
3. Kulkarni MR. Head and neck cancer burden in India. Int J Head Neck Surg. 2013; 4(1): 29- 35.
4. van der Valk MJM, Marijnen CAM, van Etten B, et al; Collaborative investigators. Compliance and tolerability of short-course radiotherapy followed by preoperative chemotherapy and surgery for high-risk rectal cancer: results of the international randomized RAPIDO-trial. Radiother Oncol. 2020;147:75-83.
5. Brunt AM , Haviland JS, Wheatley DA et al. Hypofractionated breast radiotherapy for 1 week versus 3 weeks (FAST-Forward): 5-year efficacy and late normal tissue effects results from a multicentre, non-inferiority, randomised, phase 3 trial Lancet, 395 (2020), pp. 1613-1626,
6. Bezjak A, Paulus R, Gaspar LE, et al. Safety and efficacy of a five-fraction stereotactic body radiotherapy schedule for centrally located non-small-cell lung cancer: NRG oncology/RTOG 0813 trial. J Clin Oncol. 2019;37:1316-1325.
7. Alongi F, Cozzi L, Arcangeli S, et al. Linac based SBRT for prostate cancer in 5 fractions with VMAT and flattening filter free beams: preliminary report of a phase II study. Radiat Oncol. 2013;8:171.
8. Tchelebi LT, Lehrer EJ, Trifiletti DM, Sharma NK, Gusani NJ, Crane CH, Zaorsky NG. Conventionally fractionated radiation therapy versus stereotactic body radiation therapy for locally ad-vanced pancreatic cancer (CRiSP): an international systematic review and meta-analysis. Cancer. 2020;126:2120-2131

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or above and less than 80 years.
2. Patient with high risk features: close (≤ 5mm) margin, presence of LVI or PNI, pT3-4.
3. Stage pT1-4 histological confirmed carcinoma of oral cavity with intermediate high risk feature.
4. Pathological N0 neck requiring ipsilateral neck PORT.
5. Karnofsky performance score greater or equal 70.
6. Timely delivery of PORT preferable within 6-12 weeks of surgery (additional delay of 1-3 weeks of delay beyond 12 weeks is permissible to accommodate for delayed wound healing or other logistics).
7. Written informed consent for treatment.
8. Available to attend long term follow- up.

Exclusion Criteria:

1. Pathologically positive neck disease.
2. Positive margin.
3. Patients requiring bilateral neck RT.
4. Patients that require re-irradiation for recurrent disease.
5. Previous radiotherapy to the head and neck region.
6. Any invasive malignancy within the previous 2 years (other than non melanomatous skin carcinoma or cervical carcinoma in situ).
7. Age < 18 years or > 80 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-02-29 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Severe late toxicity grade 3) at 2 year | 2 years
  Severe late toxicity > 3 or higher grade 3) at 2 year

SECONDARY OUTCOMES:
Loco-regional control rate | 2 years
  Time to an event [longitudinal assessment at 3, 6, 12, 18, 21 and 24 months
Disease free survival | 2 years
  Time to an event [longitudinal assessment at 3, 6, 12, 18, 21 and 24 months]
Overall Survival | 2 years
  Time to an event [longitudinal assessment at 3, 6, 12, 18, 21 and 24 months]
Regional recurrence at ipsilateral level IV | 2 years
  Time to an event [longitudinal assessment at 3, 6, 12, 18, 21 and 24 months]
Acute toxicity | Every week for first month
  RTOG scale
Late toxicity | 2 years
  RTOG scale [longitudinal assessment at 3, 6, 12, 18 and 24 months]
Swallowing function | 2 years
  MD Anderson Dysphagia Inventory [longitudinal assessment at 3, 6, 12, 18 and 24 months]
Quality of life EORTC QLQC30 | 2 years
  EORTC QLQC30 module [longitudinal assessment at 3, 6, 12, 18 and 24 months] The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. High score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Quality of life H&B35 | 2 years
  EORTC H&B35 module [longitudinal assessment at 3, 6, 12, 18 and 24 months]
  The head & neck cancer module incorporates seven multi-item scales that assess pain, swallowing, senses (taste and smell), speech, social eating, social contact and sexuality. There are also eleven single items. For all items and scales, high scores indicate more problems (i.e. there are no function scales in which high scores would mean better functioning). The scoring approach for the QLQ-H&N35 is identical in principle to that for the symptom scales / single items of the QLQ-C30.

CONTACTS AND LOCATIONS:
Locations (1):
- Nci, Aiims-Jhajjar, Jhajjar, Haryana, India

IPD SHARING:
Plan to Share IPD: No